CLINICAL TRIAL: NCT01832844
Title: Effects of Scan Control for Presumed Difficult Epidural Infiltrations: a Monocentric, Prospective, Randomized, Controlled, Simple Blind Trial
Brief Title: Effects of Control Scan for Presumed Difficult Epidural Infiltrations (ECHORACHIS)
Acronym: ECHORACHIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: RC13_0096
Record Dates: First submitted 2013-04-04; First posted 2013-04-16 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Sciatica
Keywords: Scan control; Epidural infiltration; visual analogue scale (VAS)
MeSH Terms: conditions — Sciatica | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group " with scan prior to infiltration " (Active Comparator)
  Interventions: Procedure: Group " with scan prior to infiltration "
- Group " without scan " (Placebo Comparator): Patients will have a "dummy" lumber spine evaluation in order to put patients in blind conditions
  Interventions: Procedure: Group " without scan "

INTERVENTIONS:
Procedure: Group " with scan prior to infiltration " — Scan will be conducted by the operator performing the gesture. He will examine the lumbar spine from L3 to S1, in longitudinal and cross sections and determine the best surgical approach. This will be defined by the largest interspinous space or better visibility of the epidural space. The depth of the epidural space will be noted. The selected stage will be marked with a skin pen to facilitate its location thereafter
  Arms: Group " with scan prior to infiltration "
Procedure: Group " without scan "
  Arms: Group " without scan "

SUMMARY:
The aim of this care protocol is to study the effects of scan to help epidural infiltration realization, in presumed difficult patients suffering from sciatica.

These scans are already performed in our Rheumatology Department but our objective is to evaluate objectively its contribution for patients and doctors.

Epidural infiltration in young patients, with an easy anatomical identification, causes generally no technical difficulties, therefore this protocol will only include patients presumed to have a difficult infiltration, that means those aged more than 60, and/or with BMI > 30 and/or suffering from scoliosis.

This study concerns patients who are hospitalized in Rheumatology Department (Hospital of Nantes) for their first epidural infiltration for treatment-resistant lombosciatica.

Patient will be randomized at Day 0, before infiltration. This latter will be performed in accordance to current practice.

Tolerance data (pain and satisfaction) will be collected just after the infiltration and eventual complications will be reported within 48 hours after infiltration.

Following treatment of lombosciatic will be realized through hospitalization, as usual.

Scan is a safe, non invasive, painless and non radiating exam. It is the extension of the musculoskeletal clinical exam and it has already changed our rheumatology practices. The investigators hope at the end of this study, that results would confirm that scan can be a help in practice to perform epidural infiltrations.

ELIGIBILITY:
Inclusion Criteria:

* Major patients hospitalized in Rheumatology Department for performing their first epidural infiltration when sciatica is resistant to medical treatment.
* Inclusion of patients older than 60 years and / or BMI superior to 30 and / or scoliosis

Exclusion Criteria:

* Refusal to participate
* History of spinal surgery
* Anticoagulant or antiplatelet
* History of spinal malformations type spina bifida
* pregnancy
* Age<18
* Patients under guardianship
* Patients participating to another clinical trial (except non interventional trials)
* Patients unable to achieve the protocol, in the judgment of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale measuring the pain during infiltration | 10min after the infiltration
  To evaluate if scan prior to epidural infiltration could improve its tolerance

SECONDARY OUTCOMES:
Infiltration evaluation: procedure time between skin passage and release of the needle | 10min after the infiltration
Infiltration evaluation: attempts number before correct positioning of needle | 10min after the infiltration
Infiltration evaluation: number of puncture sites | 10min after the infiltration
Infiltration evaluation: number of failures | 10min after the infiltration
Infiltration tolerance : VAS for pain (graduating from 0 to 10) | 48 hours
Infiltration tolerance : infiltration complications (headaches, pain at the puncture site, other) | 48 hours
Distance skin- épidural space (mm) L3-L4, L4-L5 and L5-S1 | 10min after the infiltration
Minimal interspinous distance (mm) L3-L4, L4-L5 and L5-S1 | 10min after the infiltration
Epidural space visibility L3-L4, L4-L5 and L5-S1: 0 for " no visibility ", 1 for " mild ", 2 for " good " | 10min after the infiltration
Epidural space accessibility L3-L4, L4-L5 and L5-S1 : 0 for " no visibility ", 1 for " mild ", 2 for " good " | 10min after the infiltration

CONTACTS AND LOCATIONS:
Overall Officials: Benoit LE GOFF, Doctor, Principal Investigator — Nantes University Hospital
Locations (1):
- University Hospital, Nantes, France